CLINICAL TRIAL: NCT06893757
Title: Prospective Cohort of People Starting Treatment for Tuberculosis Disease in France - ANRS 464s FrenchTB
Brief Title: Prospective Cohort of People Starting Treatment for Tuberculosis Disease in France (FrenchTB)
Acronym: FrenchTB
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Bordeaux (Other); Amiens University Hospital (Other); Centre National de la Recherche Scientifique, France (Other); Saint Antoine University Hospital (Other); University of Lyon (Other); Claude Bernard University (Other); University Hospital, Bordeaux (Other); Saint-Louis Hospital, Paris, France (Other); Centre Hospitalier Universitaire, Amiens (Other); Hôpital Jean Verdier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0464s FrenchTB; 2024-A01834-43 (Other: ID RCB)
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis
Keywords: infectious diseases; tuberculosis; clinical; social sciences; public health; Comorbidities; epidemiology; Treatment and care; Transmission; France; biobank; mycobacterial collection; cohort; prospective
MeSH Terms: conditions — Tuberculosis; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * Blood samples for the storage of whole blood, plasma, PBMCs
  * Urine samples
  * Exhaled breath condensate or exhaled breath (in a subgroup of participants)
  * Samples of other fluids or tissues depending on the investigations (body fluids, biological fluids, biopsy tissue) carried out as part of routine care and for which a sample is available (no additional sample)
  * Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- No Intervention: People starting treatment for tuberculosis disease

SUMMARY:
The French Tuberculosis Cohort is a prospective, national, multicenter, low-intervention study including subjects aged 18 years and older with tuberculosis disease for which inpatient treatment is initiated. The goal of this observational study is to follow-up and anti-tuberculosis treatment will be provided according to current French recommendations. Participants will provide sociodemographic, clinical, biological, radiological and bacteriological data at various protocol visits at 2 days, 1 and 2 weeks, 2 months, at the end of treatment, 12 and 24 months. Consenting participants will have samples collected at scheduled visits for the establishment of a biobank. This will include blood, urine, breath and hair samples. The positive mycobacterial strains will constitute a specimen bank.

DETAILED DESCRIPTION:
Main objectif:

To describe the sociodemographic, clinical, radiologic, and bacteriologic characteristics, as well as comorbidities and their impact on treatment outcomes and relapse rate up to 24 months after the start of anti-tuberculosis treatment in people with tuberculosis disease diagnosed in France.

Secondary objectives:

* Evaluate the effects of immunosuppression (HIV infection, organ transplantation, immunosuppressive treatments) on tuberculosis symptomatology, complications (including immune reconstitution inflammatory syndromes (IRIS), and drug interactions), treatment response and survival.
* Describe the characteristics of severe (meningeal, pericardial, miliary, etc.) or complicated forms of tuberculosis, including resistant tuberculosis, their management (treatment of resistant TB, use of anti-TNF, corticoids), their impact on treatment outcomes, relapse rates up to 24 months, sequelae and survival.
* Describe representations of the disease and its care, its impact on quality of life, and the effect of social determinants, situations of precariousness, health literacy, belonging to key populations (incarcerated, migrant and/or homeless people) as well as mental health disorders and addictions on compliance, experience of the disease, follow-up, and treatment outcomes.
* Describe the effect of new short-course tuberculosis treatments on adherence, disease experience, follow-up and treatment outcomes.
* Describe post-tuberculosis pulmonary sequelae, study their association with immunosuppression, pharmacological dosages, other comorbidities, tobacco and alcohol consumption, and measure physiological, structural and functional disorders, their impact on quality of life and survival.
* Study the potential diagnostic and prognostic value of new biomarkers in people with tuberculosis and the effect of exposure to anti-tuberculosis treatment on response to tuberculosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Diagnosis of tuberculosis by microbiological or clinical means, including on the basis of a pathological examination for extrapulmonary tuberculosis leading to a Compulsory Declaration (CD) and treated for less than 8 days.
* Have signed a voluntary, informed and written consent (at the latest on the day of inclusion and before any examination carried out as part of the research), or alternatively, consent from relatives in cases of tuberculous meningitis or other serious forms of tuberculosis with impaired consciousness or confusion, until the person is able to give their consent.

Exclusion Criteria:

* Presence of significant cognitive impairment that, in the opinion of the site investigator or designated person, may affect the ability to give reliable informed consent (except in the specific case of meningeal tuberculosis).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All persons included in the cohort will be followed up as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
the success of the anti-tuberculosis treatment | through treatment completion; Month 12
  Definite cure (microbiological): negative cultures (or direct examination) of respiratory specimens on two occasions during follow-up, in the last month of treatment and on an intermediate specimen, in a participant who has completed treatment and has never met the definition of treatment failure.
Success of the anti-tuberculosis treatment | through treatment completion; Month 12
  Probable cure: clinical and radiological improvement of tuberculosis-related symptoms in a participant who has completed treatment and never met the definition of treatment failure.

SECONDARY OUTCOMES:
Early microbiological response | Month 2
  Assessed by the conversion (negativation) of cultures specimens on two occasions during follow-up, in the last month of treatment and on an intermediate specimen, in a participant who has completed treatment and has never met the definition of treatment failure.
Treatment failure | Month 5
  Number of positive sputum culture
Treatment failure | Month 5
  Number of deaths directly related to tuberculosis in the year following diagnosis
Treatment failure | Month 5
  Number of interrupted treatments before the end of the planned duration and not resumed (for a reason other than a rejected tuberculosis diagnosis
Treatment failure | Month 12
  Number of treatment ongoing at 12 months because interrupted for more than two months or modified for resistance, side effects/intolerance, initial failure
Treatment failure | Month 5
  Number of transfers or loss of follow-up
Deaths | Until Month 24
  After inclusion and causes
Relapses of tuberculosis | through treatment completion until Month 24
  Positive culture of respiratory samples after the end of treatment and after cultures become negative during treatment
Relapses of tuberculosis | through treatment completion until Month 24
  Decision by the clinician to resume treatment due to suspected relapse.
Clinical and radiological post-tuberculosis respiratory sequelae and not related to another pulmonary pathology | treatment completion until Month 24
  Rate of persistent respiratory symptoms such as coughing, dyspnoea, chest pain and/or wheezing
Clinical and radiological post-tuberculosis respiratory sequelae and not related to another pulmonary pathology and/or hypoxaemia | treatment completion until Month 24
  Oxygen saturation 88% or lower and PaO2 lower 60 mmHg in ambient air at a distance from an acute episode
Clinical and radiological post-tuberculosis respiratory sequelae and not related to another Pulmonary pathology | Baseline, completion or failure treatment (up to 12 months)
  and/or impaired lung function as measured by spirometry (FEV1 or FVC <80% of the theoretical value or FEV1/FVC ratio <0.70) iv) and/or radiological sequelae defined as the persistence of pulmonary parenchymal abnormalities (nodules, cavities, reticulations, etc.). The anomalies should not be linked to an obvious cause unrelated to tuberculosis (COPD).
Functional impact and repercussions of respiratory sequelae | Baseline, Month 12, completion or failure treatment
  The he 3 components of the St Georges's Respiratory Questionnaire (SGRQ): symptoms (frequency and severity), activity (effects on and adjustment of everyday activities), and psychosocial impact. The total score has a maximum of 100 points, with values ranging from 0 to 100.
Functional impact and repercussions of respiratory sequelae | Completion treatment, Month 24
  Functional evaluation measured by the 6-minute walk test
Functional impact and repercussions of respiratory sequelae | Completion treatment (up to 12 months), Month 24
  Spirometry - FEV1/FVC ratio of greater than 0.70 and both FEV1 and FVC above 80% of the predicted value
Functional impact and repercussions of respiratory sequelae | Baseline, week 2, Month 12, completion or failure of treatment (up to 12 months), Month 24
  Pulse oximetry
Functional impact and repercussions of respiratory sequelae | Baseline, Month 2, completion or failure of treatment, Month 24
  Imaging (scanner)
Functional impact and repercussions of respiratory sequelae | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Chest X-ray2
Functional impact and repercussions of respiratory sequelae | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Other imaging for extrapulmonary involvement
Quality of life and mental health | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Psycho-trauma screening (PC-PTSD-5) - 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version.
Quality of life and mental health | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Anxiety questionnaire (GAD-7) - Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety
Quality of life and mental health | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Depression (PHQ-9) -Total scores of 5, 10, 15 and 20 represent the thresholds for mild, moderate, moderately severe and severe depression, respectively. Note: Question 9 is a single screening question on suicide risk.
Quality of life and mental health | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  EQ-5D-5L - The UI is calculated from patient scoring of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). For each dimension, participants are asked to mark between 1: 'no problems' to 5: 'unable to/extreme problems'.
Quality of life and mental health | Baseline, Day 3, Day 7
  Psycho-trauma screening (PC-PTSD-5) - 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version.
Quality of life and mental health | Baseline, Day 3, Day 7
  Hunger scale (HHS) - rating scale from 0 to 10, where 0 is painful hunger and 10 is painful fullness.
Quality of life and mental health | Completion of treatment (up to 12 months)
  Stigma scale - Responses to each item are measured on a five-point scale (ranging from zero 'strongly disagree' to four 'strongly agree'). Higher scores indicate higher levels of depression stigma.
Quality of life and mental health | Baseline, Day 3, Day 7, Month 12, completion or failure of treatment, Month 24
  Tobacco questionnaire (Fagerström) - Test for Nicotine Dependence, the three yes/no items are scored 0 (no) and 1 (yes). The three multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10.
Quality of life and mental health | Baseline, Day 3, Day 7, Month 12, completion or failure of treatment, Month 24
  Alcohol questionnaire (AUDIT-C) - scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Adherence to tuberculosis treatment | Week 2, Month 2, completion of treatment
  Psychoactive substances questionnaire (CAGE-AID) - Item responses on the CAGE are scored 0 or 1, with a higher score an indication of alcohol problems. A total score of 2 or greater is considered clinically significant. A score of 2 to 3 indicates a high index of suspicion and a score of 4 is virtually diagnostic for alcoholism.
Health literacy | Baseline, Day 3, Day 7
  Questionnaire
Screening for precariousness | Baseline, Day 3, Day 7, Month 2, Month 12
  PRECAR score
Complementary support for medical follow-up to compliance with treatment | Month 2, completion of treatment, Month 12
  Questionnaire
Only in case of TB meningitis | Baseline, Month 2, completion or failure of treatment (up to 12 months)
  Neurocognitive scores - Rankin (MR,) - Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie DE CASTRO, MD PHD, Principal Investigator — Hôpital Saint Louis Paris